CLINICAL TRIAL: NCT01461967
Title: A Single-Center, Randomized, Double-Blind, Single and Multiple Ascending-Dose, Placebo-Controlled Study to Investigate the Safety, Tolerability, Pharmacokinetics (Including the Effect of Food) and Pharmacodynamics of RO5508887 Following Oral Administration in Healthy Subjects.
Brief Title: A Study on Safety, Pharmacokinetics and Pharmacodynamics of RO5508887 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: WP25752; 2011-002053-54 (EudraCT Number)
Record Dates: First submitted 2011-10-24; First posted 2011-10-28 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteer

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Part 1a (Experimental)
  Interventions: Drug: RO5508887
- Part 1b (Placebo Comparator)
  Interventions: Drug: Placebo
- Part 2 (Experimental)
  Interventions: Drug: RO5508887

INTERVENTIONS:
Drug: Placebo — Single ascending doses
  Arms: Part 1b
Drug: RO5508887 — Single ascending doses
  Arms: Part 1a
Drug: RO5508887 — Single doses
  Arms: Part 2

SUMMARY:
This randomized, double-blind, placebo-controlled, cross-over study will assess the safety, pharmacokinetics and pharmacodynamics of RO5508887 in healthy volunteers. In Part 1, subjects will be randomized to receive single ascending doses of either RO5508887 or placebo. In Part 2, subjects will receive a single dose of RO5508887 on two occasions, with or without food. Anticipated time on study is up to 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers, 18-45 (Part 1) or 18-65 (Part 2) years of age inclusive; healthy status is defined by absence of evidence of any active or chronic disease
* Body Mass Index (BMI) 18 to 30 kg/m2 inclusive
* Male subjects must use a barrier method of contraception for the duration of the study and for 30 days after the last dose

Exclusion Criteria:

* Suspicion of regular consumption of drugs of abuse
* Regular smoker (>5 cigarettes, >1 pipeful or >1 cigar per day)
* Positive for hepatitis B, hepatitis C or HIV infection
* History of hypersensitivity or severe drug reaction
* Participation in an investigational drug or device study within three months before the first drug administration

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2011-09; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Safety/tolerability: Incidence of adverse events | up to approximately 8 weeks

SECONDARY OUTCOMES:
Pharmacokinetics: Plasma concentrations of RO5508887 | predose, 1.5, 3, 4, 4.5, 5, 5.5, 6, 7, 8, 12, 24, 48, 72, 96, 144 hours post-dose
Pharmacodynamics: Urine levels of RO5508887 | predose to 72 hours post-dose
Pharmacodynamics: Plasma levels of markers of amyloid deposition (Abeta1-40/Abeta1-42) | predose, 1.5, 3, 4, 4.5, 5, 5.5, 6, 7, 8, 12, 24, 48, 72, 96, 144 hours post-dose
Effect of food on pharmacokinetics (plasma concentrations) of a single dose of RO5508887 | predose, 1.5, 3, 4, 4.5, 5, 5.5, 6, 7, 8, 12, 24, 36, 48, 60, 72 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Strasbourg, France